CLINICAL TRIAL: NCT02741258
Title: Mepitel Film vs Standard of Care for the Radiotherapy Prevention and Cutaneous Toxicity in Patients With Post-surgery Breast Cancer
Brief Title: Mepitel Film Treatment for the Prevention and Cutaneous Toxicity Due to Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dario Valcarenghi (Other)
Responsible Party: Sponsor-Investigator, Dario Valcarenghi, Clinical Research Nurse, Oncology Institute of Southern Switzerland
Organization: Oncology Institute of Southern Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-INF-001
Record Dates: First submitted 2016-03-15; First posted 2016-04-18 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Post-surgery Radiotherapy
MeSH Terms: interventions — Skin Cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepitel Film (Experimental): Mepitel film will be placed on the patients' skin just before the start of the radiotherapy and will be replaced once a week until the end of the radiotherapy. In case of skin toxicities mepitel film will be placed until resolution of the toxicities. In case of new skin toxicities appearance the patient will be retreated with Mepitel.
  Interventions: Device: Mepitel Film
- Excipial U hydrolotion, Flammazin skin cream (Active Comparator): Patients will be treated with aqueous (Excipial U hydrolotion) or antiseptic (Flammazine or Ialugen Plus) cream in case of skin erythema due to radiotherapy. In case of new skin toxicities appearance the patient will be retreated with standard of care treatment.
  Interventions: Drug: skin cream

INTERVENTIONS:
Device: Mepitel Film — Placement of Mepitel Film to prevent skin toxicity
  Arms: Mepitel Film
Drug: skin cream — cream to treat skin erythema due to radiotherapy
  Other Names: Excipial U hydrolotion, Flammazin
  Arms: Excipial U hydrolotion, Flammazin skin cream

SUMMARY:
This is a randomized study, mepitel vs standard of care for the prevention and skin toxicity due to radiotherapy in patients with post-surgery breast cancer.

Mepitel film will be placed on the skin of the patients just before the start of the radiotherapy and will be replaced once a week until the end of the radiotherapy. In case of skin toxicities mepitel film will be placed until resolution of toxicities.

DETAILED DESCRIPTION:
For patients randomized in the mepitel arm:

Mepitel film will be placed on the patients' skin just before the start of the radiotherapy and will be replaced once a week until the end of the radiotherapy. In case of skin toxicities mepitel film will be placed until resolution of the toxicities. In case of new skin toxicities appearance the patient will be retreated with mepitel.

For patients randomized in the standard of treatment arm:

Patients will be treated with aqueous (Excipial U hydrolotion) or antiseptic (Flammazine o Ialugen Plus) cream in case of skin erythema. In case of new skin toxicities appearance the patient will be retreated with standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer treated with conservative surgery who need radiotherapy treatment
* capability and willness to participate to the study
* informed consent form signature

Exclusion Criteria:

* contraindication to the correct placement of the Mepitel Film
* previous breast radiation treatment
* participating in other clinical trials
* previous breast reconstruction
* concomitant treatment with antiblastic chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mepitel Film efficacy in treating skin toxicity evaluatet with Common Terminology Criteria for Adverse Events (CTCAE) | one week after start of radiotherapy
  Common Terminology Criteria for Adverse Events (CTCAE) V.4 will be used to evaluate the toxicity

SECONDARY OUTCOMES:
Time for the skin toxicity appearance and resolution | one week after start of radiotherapy
Severity of the chronic skin toxicity | one week after start of radiotherapy
  Common Terminology Criteria for Adverse Events (CTCAE) v.4

CONTACTS AND LOCATIONS:
Overall Officials: Dario Valcarenghi, Study Chair — Oncology Institute of Southern Switzerland
Locations (2):
- Switzerland (2):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Institut für Radiotherapie Klinik Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No
not foreseen